CLINICAL TRIAL: NCT06338813
Title: Comparison of the Kron Technique and Digital Manometry for Intra-Abdominal Pressure Measurement in Emergency Department Patients Diagnosed With Ileus
Brief Title: Digital Manometry for Intra-Abdominal Pressure Measurement in Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cagdas Yildirim, MD, Asistant Professor, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: Merve Unutmaz
Record Dates: First submitted 2024-03-19; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Kron Technique (No Intervention): Intraabdominal pressure measurement with Kron Technique
- Digital Manometry (Active Comparator): Intraabdominal pressure measurement with Digital Manometry
  Interventions: Device: Digital Manometry

INTERVENTIONS:
Device: Digital Manometry — The "Compass Lumbar Puncture Pressure Transducer" (Mirador Biomedical, Seattle, WA, USA) was used as a digital manometer. After the bladder was completely emptied, the catheter was clamped again. 25 cc of sterile saline was injected into the bladder through the urine sample port. The digital manometer was connected to the urine sample port. The IAP value in cmH2O on the digital screen of the device was noted.
  Arms: Digital Manometry

SUMMARY:
Although many measurement techniques have been tried for intra-abdominal pressure, the Kron technique is currently the gold standard method. However, the search for other methods continues due to its long application time, the need for more equipment, and impracticality. Consequently, the investigators sought to investigate a quicker and more accessible method suitable for successful intra-abdominal pressure measurement in the emergency department. This study aimed to compare intra-abdominal pressure measurements in patients diagnosed with ileus using a digital manometer and the Kron Technique.

DETAILED DESCRIPTION:
Before the start of the study, the Kron Technique and IAP measurement with a digital manometer were demonstrated both didactically and practically to 4th year Emergency Medicine residents. It was ensured that any two of these residents were continuously present on the monthly duty roster. When a patient who met the inclusion criteria presented to the emergency department, the residents were separately invited to the bedside for measurements by the attending physician without each other's knowledge. After the attending physician obtained information about the patient, the exclusion criteria were evaluated. After the patient was deemed eligible, the attending physician explained the application and the study to the patient in detail. Informed consent was obtained from the patients both verbally and in written. Demographic information (age, gender) and medical history were recorded.

Measurements were performed with the patient in the supine position. A transurethral Foley catheter (16 Fr) was inserted by the attending physician under sterile conditions. First, IAP was measured using the 'Kron technique.' The connection hose of the urine collection container was attached to the Foley catheter. The hose was clamped after the urine in the bladder was completely emptied. A sterile three-way tap was attached to the urine sample port in the connection hose. From the three-way tap, 25 ml of sterile saline was injected into the bladder with a syringe. Subsequently, one end of the transducer interconnection cable was connected to the three-way tap, and the other end was connected to the bedside monitor (GE B40 V3 bedside monitor, Germany). Subsequently, pressure adjustments were reset on the monitor, and IAP was recorded in mmHg. After this measurement, a digital manometer was used. This measurement was performed by the second resident. The "Compass Lumbar Puncture Pressure Transducer" (Mirador Biomedical, Seattle, WA, USA) was used as a digital manometer (Figure 2). After the bladder was completely emptied, the catheter was clamped again. 25 cc of sterile saline was injected into the bladder through the urine sample port. The digital manometer was connected to the urine sample port. The IAP value in cmH2O on the digital screen of the device was noted. The IAP measurement value recorded in cmH2O was converted to mmHg using the equation "1 cmH2O = 0.7355 mmHg." During the measurements, the patient's treatment plan was not interrupted.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* Diagnosis of ileus was confirmed by radiological imaging (radiography and Computed Tomography)

Exclusion Criteria:

* Patients who underwent any decompressive procedure before the measurement (Nasogastric catheter, enema)

  * Patients who could not be urine catheterized
  * Patients who could not be placed in the supine position (advanced heart failure, kyphosis, etc.)
  * Uncooperative patients (Alzheimer's, dementia, mental retardation, etc.)
  * Patients with morbid obesity (body mass index > 40 kg/m2), ascites, or pregnancy
  * Patients who have undergone bladder surgery
  * Patients with neurogenic bladder

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Digital manometer measuring for Intraabdominal Pressure | 30 minutes
  Compare the Kron technique, which is a more complex method but considered the gold standard, with Intraabdominal Pressure measurement using a digital manometer

CONTACTS AND LOCATIONS:
Overall Officials: Çağdaş Yıldırım, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)